CLINICAL TRIAL: NCT05807971
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of ATH-063 in Healthy Subjects
Brief Title: Assessment of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ATH-063 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athos Therapeutics Inc (Industry)
Collaborators: Syneos Health (Other); Athos Therapeutics Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATH-001
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Autoimmune Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Cohorts (4 each) within the SAD and MAD part will be dosed sequentially in an ascending fashion.
  MAD cohorts and FE cohort will be dosed in parallel after the completion of the SAD Cohorts.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be double-blinded. The subjects and the clinical personnel involved in the collection, monitoring, revision, or evaluation of AEs, or personnel who could have an impact on the outcome of the study will be blinded with respect to the subject's treatment assignment (ATH-063 or placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SAD cohort (Experimental): SAD cohorts 1-4. Subjects in each cohort will be randomized to receive a single oral dose of ATH-063 (capsule) under fasting conditions at the planned dose levels.
  Interventions: Drug: ATH-063
- MAD Cohort (Experimental): MAD cohorts 1-4. Subjects in each cohort will be randomized to receive multiple oral doses of ATH-063 (Capsule) under fasting conditions once daily (QD) for 10 consecutive days at planned dose levels.
  Interventions: Drug: ATH-063
- Food Effect (Experimental): An intermediary dose level that has already been administered in this study will be selected for the food-effect evaluation based on the available PK and safety data. This will be conducted under fasting and fed conditions.
  Interventions: Drug: ATH-063
- SAD cohort (Placebo) (Placebo Comparator): SAD cohorts 1-4. Subjects in each cohort will be randomized to receive a single oral dose of placebo (Capsule identical to active ATH-063) under fasting conditions at the planned dose levels.
  Interventions: Drug: Placebo
- MAD cohort (Placebo) (Placebo Comparator): MAD cohorts 1-4. Subjects in each cohort will be randomized to receive multiple oral doses of placebo (Capsule identical to active ATH-063) under fasting conditions once daily (QD) for 10 consecutive days at planned dose levels.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATH-063 — 12.5 and 50 mg Capsules, anticipated dose range to be from 25 to 250 mg.
  Arms: Food Effect; MAD Cohort; SAD cohort
Drug: Placebo — Identical capsule to the drug without the active ingredient.
  Arms: MAD cohort (Placebo); SAD cohort (Placebo)

SUMMARY:
The goal of this clinical trial is to test the ATH-063 drug (single and multiple doses) in Healthy Subjects. The clinical trial aims to evaluate the below.

1. Safety of the drug
2. Tolerability of the drug
3. Pharmacokinetics (PK) (how the human body affects the drug)
4. Pharmacodynamics (PD) (how the drug affects the human body)

This will be a single center, Phase 1, First-In-Human, Randomized, Double-Blind (neither the subjects nor the experimenters know which subjects are in the test and control groups), Placebo (a look-alike substance that contains no active drug) - Controlled Study.

DETAILED DESCRIPTION:
Primary Objective of this study will be to evaluate the safety and tolerability of ATH-063 following oral administration of single and multiple ascending doses (SAD/MAD) in healthy subjects.

This is a single center, Phase 1, Randomized, Double-blind, Placebo controlled, sequential SAD/MAD study, with a food-effect arm. The study will be divided into three parts:

* SAD cohorts
* MAD cohorts
* Food-effect (FE) cohort

MAD and FE cohorts will be dosed in parallel after the completion of the SAD Cohorts

SAD Part:

1. Consist of at least 4 cohorts (1 cohort per dose level).
2. Each cohort will include approximately 8 participants (6 participants receiving the active and 2 participants receiving the placebo).
3. A staggered dosing schedule will be used for dosing of each cohort (under fasting conditions)

MAD Part:

1. Consist of up to 4 cohorts (1 cohort per dose level).
2. Each cohort will include approximately 8 participants (6 participants receiving the active and 2 participants receiving the placebo).
3. The cohorts will be dosed sequentially in an ascending fashion.
4. The dose of MAD cohorts is dependent on the available safety, tolerability, and PK data from the SAD part and available safety, tolerability, and PK data from dosed MAD cohorts.

Food-effect Part:

1. Approximately twelve (12) participants will be randomized in a 1:1 ratio to one of two treatment sequences (fast-fed/fed-fast) with 6 participants per treatment sequence.
2. The selection of the dose to be administered in the food effect part will depend on the results of the SAD part following the review of safety, tolerability and PK data of the SAD cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening) or social smoker (smokers with 1-5 cigarettes a week), AND with a negative urine cotinine test at check-in, ≥18 and ≤55 years of age, with BMI >18.5 and <32.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females and a maximum weight of 120 kg.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to study drug administration.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease. A history of migraines, childhood asthma, or non-hospitalized depression would not be considered clinically significant.
3. Female participants of non-childbearing potential must be:

   1. post-menopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with confirmation by documented follicle-stimulating hormone (FSH) levels ≥ 40 mIU/mL; or
   2. surgically sterile (bilateral oophorectomy, bilateral salpingectomy, hysterectomy, or tubal ligation) at least 3 months prior to dosing.
4. Sexually active females of childbearing potential and non-sterile males must be willing to use an acceptable contraceptive method throughout the study as detailed in section 8.1.
5. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination.
2. Clinically significant abnormal laboratory test results or positive serology test results for HBsAg, HCV antibody, or HIV antigen and antibody, at screening.
3. Positive pregnancy test or lactating female subject
4. Positive urine drug screen, urine cotinine test, or alcohol breath test (one repeat is allowed).
5. History of significant allergic reactions (e.g., anaphylactic reaction, hypersensitivity, angioedema) to any drug.
6. Clinically significant ECG abnormalities or vital signs abnormalities (systolic BP lower than 90 or over 160 mmHg, diastolic BP lower than 50 or over 95 mmHg, HR less than 45 or over 100 bpm, or RR less than 12 or over 22 bpm) at screening.
7. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
8. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 375 mL of beer 3.5%, 100 mL of wine 13.5%, or 45 mL of distilled alcohol 40%). Low risk level = 10 unites per week for men and women.
9. Use of medications for the timeframes specified below, with the exception of hormonal contraceptives and medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

   1. depot injection or implant within 3 months prior to the first dosing;
   2. live attenuated vaccines within 1 month prior to the first dosing;
   3. any drug known to induce or inhibit hepatic drug metabolism, including St. John's wort, within 30 days prior to the first dosing;
   4. prescription medications within 14 days prior to the first dosing;
   5. any other vaccine, including COVID-19 vaccine, within 14 days prior to the first dosing;
   6. over-the-counter (OTC) medications and natural health products (including herbal remedies such as, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first dosing, with the exception of the occasional use of paracetamol (up to 2 g daily).
10. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days or 5 x T1/2 whichever is longer prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days or 5 x T1/2 whichever is longer prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
11. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
12. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ATH-063 following oral administration of single and multiple ascending doses in healthy participants. | SAD: Up to 15 ± 1 day, MAD: Up to 24 ± 1 day, FE: Up to 14 ± 1 day
  Number of participants with serious and other non-serious adverse events

SECONDARY OUTCOMES:
Pharmacokinetic assessment 1 | SAD: Up to 15 ± 1 day, MAD: Up to 24 ± 1 day, FE: Up to 14 ± 1 day
  AUC0-t (Area under the plasma concentration-time curve)
Pharmacokinetic assessment 2 | SAD: Up to 15 ± 1 day, MAD: Up to 24 ± 1 day, FE: Up to 14 ± 1 day
  AUC0-inf (AUC curve to infinite time)
Pharmacokinetic assessment 3 | SAD: Up to 15 ± 1 day, MAD: Up to 24 ± 1 day, FE: Up to 14 ± 1 day
  Cmax (Maximum plasma concentration)
Pharmacokinetic assessment 4 | SAD: Up to 15 ± 1 day, MAD: Up to 24 ± 1 day, FE: Up to 14 ± 1 day
  Tmax (Time to maximum plasma concentration (Cmax)
Pharmacokinetic assessment 5 | SAD: Up to 15 ± 1 day, MAD: Up to 24 ± 1 day, FE: Up to 14 ± 1 day
  Residual area
Pharmacokinetic assessment 6 | SAD: Up to 15 ± 1 day, MAD: Up to 24 ± 1 day, FE: Up to 14 ± 1 day
  T½ el (Half Life)
Pharmacokinetic assessment 7 | SAD: Up to 15 ± 1 day, MAD: Up to 24 ± 1 day, FE: Up to 14 ± 1 day
  Kel (Elimination rate constant)
Pharmacokinetic assessment 8 | SAD: Up to 15 ± 1 day, FE: Up to 14 ± 1 day
  Cl/F (Oral Clearance)
Pharmacokinetic assessment 9 | MAD: Up to 24 ± 1 day
  Clss/F (Oral Clearance-steady state)
Pharmacokinetic assessment 10 | SAD: Up to 15 ± 1 day, FE: Up to 14 ± 1 day
  Vz/F (Apparent volume of distribution)
Pharmacokinetic assessment 11 | MAD: Up to 24 ± 1 day
  AUC0-24 (area under the plasma concentration-time curve over the last 24-h dosing interval)
Pharmacokinetic assessment 12 | MAD: Up to 24 ± 1 day
  AUC0-tau (area under the curve to the end of the dosing period)
Pharmacokinetic assessment 13 | MAD: Up to 24 ± 1 day
  Cmax ss (Maximum plasma concentration at steady state)
Pharmacokinetic assessment 14 | MAD: Up to 24 ± 1 day
  Tmax ss (Time to steady state Cmax)
Pharmacokinetic assessment 15 | MAD: Up to 24 ± 1 day
  Cmin ss (Minimum drug concentration at steady-state)
Pharmacokinetic assessment 16 | MAD: Up to 24 ± 1 day
  Vz ss/F (Apparent volume of distribution at steady state)
Pharmacokinetic assessment 17 | FE: Up to 14 ± 1 day
  Tlag (Lag time)

OTHER OUTCOMES:
Pharmacodynamic assessment 1 | MAD: Up to 24 ± 1 day
  change from baseline in T-regulatory cells immunophenotype
Pharmacodynamic assessment 2 | MAD: Up to 24 ± 1 day
  change from baseline in T-regulatory cells H3K9 methylation status
Pharmacodynamic assessment 3 | MAD: Up to 24 ± 1 day
  change from baseline in plasma proteomic signature
Pharmacodynamic assessment 4 | MAD: Up to 24 ± 1 day
  change from baseline in stool microbiome signature

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Farinola, B.Sc (Biomed. Sci.),BMBS,FRACP, Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No